CLINICAL TRIAL: NCT07113704
Title: Fundus-First Laparoscopic Cholecystectomy in Difficult Gallbladders: A Retrospective Cross-Sectional Study on a Safe Alternative to Avoid Conversion
Brief Title: Fundus-First Laparoscopic Cholecystectomy in Difficult Gallbladders: A Safe Alternative Technique
Status: Completed | Type: Observational
Sponsor: KANAN ISMAYILZADA, MD (Other)
Responsible Party: Sponsor-Investigator, KANAN ISMAYILZADA, MD, General Surgeon, Medicana Ataşehir International Hospital
Organization: Medicana Ataşehir International Hospital (Other)
Other Study IDs: FFLC2025AMSUKI
Record Dates: First submitted 2025-07-25; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cholelithiasis
Keywords: fundus-first laparoscopic cholecystectomy; difficult cholecystectomy; Cross-sectional study; General surgery; Laparoscopic cholecystectomy; Tertiary care hospital
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Laparoscopic Cholecystectomy: Patients who underwent standard laparoscopic cholecystectomy, starting dissection at Calot's triangle. This technique served as the comparator for assessing safety and conversion rates relative to the fundus-first approach.
  Interventions: Procedure: Conventional Laparoscopic Cholecystectomy
- Fundus-First Laparoscopic Cholecystectomy: Patients with difficult gallbladders (Nassar Grade 3-4) who underwent laparoscopic cholecystectomy using the fundus-first technique. This approach involved starting dissection at the gallbladder fundus and proceeding retrogradely toward Calot's triangle to improve safety in complex cases.
  Interventions: Procedure: Fundus-First Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Conventional Laparoscopic Cholecystectomy — Standard laparoscopic cholecystectomy technique starting at Calot's triangle. Used as the comparator group in this study.
  Other Names: Antegrade Laparoscopic Cholecystectomy
  Groups: Conventional Laparoscopic Cholecystectomy
Procedure: Fundus-First Laparoscopic Cholecystectomy — Laparoscopic cholecystectomy technique initiated at the gallbladder fundus and carried out retrogradely toward Calot's triangle. This method was applied to difficult gallbladders (Nassar Grade 3-4) to improve operative safety and avoid conversion to open surgery.
  Other Names: Retrograde laparoscopic cholecystectomy
  Groups: Fundus-First Laparoscopic Cholecystectomy

SUMMARY:
This retrospective cross-sectional study evaluated the safety and effectiveness of the fundus-first laparoscopic cholecystectomy (FFLC) technique in patients with difficult gallbladders. A total of 124 patients who underwent FFLC between 2023 and 2024 were reviewed. The study assessed operative time, intraoperative complications, conversion rates, and postoperative outcomes. The results suggest that FFLC is a safe and feasible approach that can reduce the need for conversion to open surgery in complex cases. The study was conducted at a private hospital in Istanbul, Turkey

DETAILED DESCRIPTION:
This retrospective study was conducted at a private healthcare institution without a formal IRB. All patient data were anonymised before analysis, and written informed consent was obtained from all patients for the academic use of their clinical data

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic cholecystectomy at the study center between January 2023 and March 2024
* Patients diagnosed with difficult gallbladder (Nassar Grade 3-4)
* Age ≥ 18 years
* Complete clinical data available for analysis

Exclusion Criteria:

* Patients with incomplete medical records
* Patients undergoing open cholecystectomy from the beginning
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included adult patients (≥18 years) who underwent laparoscopic cholecystectomy for difficult gallbladder (Nassar grade 3-4) at a single tertiary care center between January 2023 and March 2024.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Conversion Rate to Open Surgery | Intraoperative (during surgery)
  Rate of conversion from laparoscopic to open cholecystectomy in each group. Measured as number and percentage of patients converted.

SECONDARY OUTCOMES:
Operative Time | Intraoperative (during surgery)
  Total operative time measured in minutes from skin incision to closure. Comparison between the fundus-first and conventional laparoscopic cholecystectomy groups.
Postoperative Complication Rate | Within 30 days postoperatively
  Includes complications such as wound infection, bile leak, abscess, or any adverse event requiring medical or surgical intervention. Compared between groups
Length of Hospital Stay | Postoperative hospitalization
  Number of days from surgery to discharge. Mean values will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: KANAN ISMAYILZADA, MD, Principal Investigator — Medicana Ataşehir International Hospital, ISTANBUL.TURKEY
Locations (1):
- Medicana Ataşehir International Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study is retrospective in nature, and no plans have been made to share individual participant data with other researchers.

DOCUMENTS (1):
  • Study Protocol (2025-08-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT07113704/Prot_000.pdf